CLINICAL TRIAL: NCT05903456
Title: Icaritin Soft Capsule Combined With Lenvatinib and Transcatheter Arterial Chemoembolization（TACE） for the Treatment of Hepatocellular Carcinomaunresectable, Non-metastatic Hepatocellular Carcinoma
Brief Title: Icaritin Soft Capsule Combined With Lenvatinib and TACE for the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Guoliang Shao, Chief Physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2022-802
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Icaritin soft capsules;TACE; lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Drug Delivery Systems

STUDY DESIGN:
Masking Description: NO masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE +lenvatinib+Icaritin soft capsules (Experimental): Trial drug Lenvatinib, 8mg (2 tablets for patients weighing less than 60kg), or 12mg (3 tablets for patients weighing more than 60kg), once daily. Icariin Soft Capsules 1200 mg/d (6 tablets in two doses) should be swallowed with warm water within 30 minutes after meal. Take lenvatinib and Icaritin soft capsules 3 to 5 days after TACE. Until the disease progresses or the patient becomes intolerant.
  Interventions: Procedure: TACE（transcatheter arterial chemoembolization）; Drug: lenvatinib; Drug: Icaritin soft capsules

INTERVENTIONS:
Procedure: TACE（transcatheter arterial chemoembolization） — TACE treatment is strictly in accordance with the Chinese guidelines for clinical practice of transcatheter arterial chemoembolization (TACE) for hepatocellular carcinoma (2018 Edition).
  The patients with HCC were selected according to the inclusion criteria (referring to the conditions of the subjects). The subjects who met the inclusion criteria could enter the study after they signed the informed consent. 4-6 weeks after the first TACE treatment, the resectability criteria were evaluated. If not, the next cycle of TACE treatment was carried out. The general principle is to reduce the number of interventional treatment and extend the interval of interventional operation as far as possible under the condition of controlling the tumor and the survival of patients with tumor.
Drug: lenvatinib — Ronvastinib is an orally administered multi-receptor tyrosine kinase (RTK) inhibitor that selectively inhibits the kinase activity of vascular endothelial growth factor (VEGF) receptors, such as VEGF-1, VEGF-2, and VEGF-3, in addition to inhibiting other pro-angiogenic and oncogenic signaling pathways associated with tumor proliferation ，has been approved as a first-line treatment for liver cancer
  Other Names: target drug
Drug: Icaritin soft capsules — Icaritin soft capsule is a flavonoid compound extracted from traditional Chinese medicinal materials. It is a new type of small molecule immunomodulator. It is a 1.2 class of innovative Chinese medicine with global independent intellectual property rights. By inhibiting inflammatory signaling pathway and reducing the release of inflammatory factors, the immune microenvironment can be regulated to play an anti-tumor role. At present, it has been approved for first-line treatment of advanced liver cancer, with good efficacy and safety.
  Other Names: Small molecule immunomodulator

SUMMARY:
The investigators design a phase II clinical study to explore the efficacy and safety of Transarterial Chemoembolization (TACE) + Lenvatinib + Icaritin soft capsules in patients with Unresectable, non-metastatic hepatocellular carcinoma and to analyze potential biomarkers of therapeutic response.

DETAILED DESCRIPTION:
This is a single-center, open-label, prospective, non-randomized clinical trial. We adopted the prospective cohort study to explore the safety and efficacy of Transarterial Chemoembolization (TACE) + Lenvatinib + Icaritin soft capsules in the patients with Unresectable, non-metastatic hepatocellular carcinoma.

It is estimated that 20 patients who met the study criteria will be enrolled in Zhejiang Cancer Hospital. The investigators will follow up and collect subjects' data monthly to evaluate the efficacy and safety of treatment, including overall survival and time to progression. Multi-omics data analysis will be used to find potential biomarkers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80;
2. Patients with histological/cytological confirmed hepatocellular carcinoma.
3. HCC patients eligible for China liver cancer staging (CNLC) Stage IIIa, which cannot be resectable, are not suitable for radical treatment.
4. According to the RECIST v1.1 standard, there must be at least one measurable lesion on the upper abdominal enhanced CT or MRI.
5. Child-Pugh grade A or B;
6. ECOG physical condition score is 0 or 1;
7. Suitable for the indications of TACE surgery and chemotherapy drugs prescribed in advance by the research center, without any contraindications.
8. Regular antiviral therapy should be given if HBV or HCV infection is present.
9. Life expectancy is more than 3 months
10. Able to swallow and absorb oral tablets;
11. Appropriate organ function with the following laboratory test values obtained within 7 days prior to therapeutic use:
12. (hemoglobin value ≥80g/L, neutrophil count ≥2.5×109/L, platelet count ≥75×109/L, serum total bilirubin ≤2× upper limit of normal (UNL), aspartic transferase ≤2×UNL, alanine transferase ≤3×UNL, serum creatinine ≤1.5×UNL)
13. Manageable blood pressure
14. Women of childbearing age must already be using reliable contraception or have had a negative pregnancy test (serum or urine) within 7 days prior to enrollment and be willing to use an effective method of contraception during the trial period and within 2 months after the last drug administration. Male subjects whose partners are women of childbearing age should use effective methods of contraception during the trial period and within 2 months after the last dose;
15. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Formation of portal vein main cancer thrombus or extensive cancer thrombus.
2. HCC was treated with local treatment of existing lesions (e.g., TACE, ablation, particle, TARE, hepatic arterial infusion chemotherapy, or radiotherapy).
3. Patients who have previously received targeted or immunoreactive anti-tumor therapy for HCC and chemotherapy need to be desensitized for more than one month.
4. Subjects were unable to perform enhanced CT or MRI scans of the liver.
5. Have a history of liver transplantation or are currently candidates for liver transplantation.
6. Patients at high risk for esophageal or gastric variceal bleeding or unproven severe variceal bleeding within the last 3 months.
7. Have bleeding or thrombotic disease or are receiving thrombolytic therapy
8. Study clinically significant hemoptysis or tumor hemorrhage of any cause within 2 weeks prior to initial administration of the intervention.
9. Study of significant cardiovascular impairment in the 12 months prior to initial administration, such as a history of congestive heart failure above NYHA Grade II (Appendix 12), unstable angina, myocardial infarction or cerebrovascular stroke, or arrhythmias associated with hemodynamic instability.
10. There was clinically significant ascites on physical examination, which could not be controlled by drugs.
11. Known to be allergic to any component of icartin soft capsules and lenvatinib preparation.
12. Pregnant or lactating female patients.
13. Other conditions in which participation in the study is not appropriate according to the investigator's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 48 weeks
  It was defined as the percentage of patients with complete response (CR) and partial response (PR) in all patients, and the treatment response was based on the modified response evaluation criteria in solid tumors (recist1.1)

SECONDARY OUTCOMES:
progression-free survival | 96 weeks
  It was defined as the time from successful hepatectomy to recurrence. Patients who withdraw or lose follow-up will be treated as deletion
Overall Survival | 96 weeks
  It was defined as the time from the beginning of treatment to death from any cause throughout the trial. Patients who dropped out or lost follow-up will be treated as deletion, and the known last survival date will be regarded as the last survival time. Patients who survived at the end of the study will also be treated as deletions, and the last known date of survival will be taken as the final survival time
Disease Control Rate | 48 weeks
  It was defined as the Proportion of all subjects receiving study therapy who rated complete response (CR), partial response (PR), and stable disease (SD) as best overall response according to RECIST 1.1 criteria.
Duration of Response | up to 48 weeks
  It was defined as the period from the date when tumor response was first recorded (as measured by RECIST 1.1 criteria) to the date when objective tumor progression was first recorded (as measured by RECIST 1.1 criteria) or the date of death from any cause.
adverse event | 96 weekes
  The incidence, severity, and serious adverse events associated with medication use were determined by NCI CTCAE v5.0 standards

IPD SHARING:
Plan to Share IPD: No